CLINICAL TRIAL: NCT06466408
Title: Exploring the Impact of Fruit and Vegetable Enzyme Supplementation on Aerobic Performance and Lactate Response in the Elderly Following High-Intensity Interval Exercise Combine Exergaming: Randomized Experimental Matched-Pair Study
Brief Title: Effect of Vegetable and Fruit Enzyme Supplementation on Muscle Activation, Aerobic Capacity, and Blood Biochemical Parameters After High-Intensity Interval Exercise: Feasibility Study of Exercise Design With Exergaming
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shu-Cheng Lin (Other)
Responsible Party: Sponsor-Investigator, Shu-Cheng Lin, Assistant Professor, Tainan University of Technology
Organization: Tainan University of Technology (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NCKU HREC-E-112-419-2
Record Dates: First submitted 2024-05-18; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Overtraining Syndrome
MeSH Terms: conditions — Overtraining Syndrome

STUDY DESIGN:
Intervention Model Description: groups -enzyme and -placebo
Who Masked: Participant
Masking Description: groups -enzyme and -placebo single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- enzyme group (Experimental): enzyme group consumed 30 mL of vegetable and fruit enzymes (The contents include needle-leaf cherries, cherries, apples, cranberries, blackberries, black currants, blueberries, beets, broccoli, cabbage, carrots, Concord grapes, cranberries, elderberries, kale, oranges, peaches, papayas, parsley, pineapples, raspberries, red currants, spinach, and tomatoes, etc.)(Enzyme Village, Chiayi, Taiwan) mixed with 150 mL of water twice a day (at breakfast and dinner) for 14 consecutive days.
  Interventions: Dietary Supplement: Supplementation Protocol; Diagnostic Test: Blood Lactate Test; Diagnostic Test: Training Impulse; Diagnostic Test: Exergaming HIIE Test
- placebo group (Placebo Comparator): The placebo group followed the same protocol but consumed malt syrup (Amazon, USA) mixed with 150 mL of water twice a day (at breakfast and dinner) for 14 consecutive days.
  Interventions: Dietary Supplement: Supplementation Protocol; Diagnostic Test: Blood Lactate Test; Diagnostic Test: Training Impulse; Diagnostic Test: Exergaming HIIE Test

INTERVENTIONS:
Dietary Supplement: Supplementation Protocol — After the pre-test, the enzyme group consumed 30 mL of vegetable and fruit enzymes (The contents include needle-leaf cherries, cherries, apples, cranberries, blackberries, black currants, blueberries, beets, broccoli, cabbage, carrots, Concord grapes, cranberries, elderberries, kale, oranges, peaches, papayas, parsley, pineapples, raspberries, red currants, spinach, and tomatoes, etc.)(Enzyme Village, Chiayi, Taiwan) mixed with 150 mL of water twice a day (at breakfast and dinner) for 14 consecutive days. The placebo group followed the same protocol but consumed malt syrup (Amazon, USA) instead until the end of the study. Participants returned to the laboratory each morning to receive the daily supplement, which was administered on-site. Following supplementation, participants reported their dinner intake to the researchers, ensuring compliance with the prescribed supplementation regimen.
Diagnostic Test: Blood Lactate Test — The blood lactate was measured at five time points: before exercise, after the fourth and eighth bouts of exercise, and at 5 and 10 minutes after exercise. The blood lactate were analyzed using a Biosen Cline blood analysis system (EKF-diagnostic, Germany). Capillary blood samples of 10 μL were collected and added to red blood cell lysis reagent and stored at low temperature until analyzed. Prior to analysis, instrument standardization and test calibration were performed, and the coefficient of variation was determined to be ≤1.5%. The detection range for blood lactate was 0.5-40 mM
Diagnostic Test: Training Impulse — In this study, the exercise load was represented by the TRIMP [32], which is calculated as the product of exercise intensity and duration. To accommodate the convenience of the experiment, two different TRIMP calculation methods were used, including % HRmax (objective) and RPE (subjective). At the end of each exercise bout (8 bouts in total) and during the recovery period before the next bout (7 bouts in total), participants were asked to report their RPE, and their heart rate was recorded. This process was repeated 8 times.
Diagnostic Test: Exergaming HIIE Test — The sensor system utilized two Nintendo controllers: one mounted on the exercise ring and the other secured to the participant's thigh to enhance gameplay interaction. Through the Ring-Con, participants engaged in diverse physical activities such as weightlifting, yoga, and aerobic exercises. The fitness ring sensor accurately captures and integrates players' movements into the game. The gameplay involves unlocking levels and engaging in fitness challenges that are achieved through actual physical activities. It offers a wide range of exercise routines targeting various muscle groups and provides engaging gaming challenges. The exercise protocol included eight sets of 20-second high-effort exercises, interspersed with 30-second rest intervals, totaling 370 seconds of active exercise time. Specifically, the fitness game mode used was the Adventure Mode in 'Ring Fit Adventure,' comprising exercises targeting the pectoralis major, latissimus dorsi, deltoids, and quadriceps muscles.

SUMMARY:
This study explores the effectiveness of fruit and vegetable enzyme supplementation in reducing fatigue and enhancing aerobic capacity in elderly individuals after engaging in high-intensity interval exercise (HIIE) through exergaming. Sixteen elderly female participants were divided into two groups based on pre-test lactate levels: an enzyme group and a placebo group, to ensure comparability. They performed HIIE using Nintendo Switch Ring Fit Adventure, completing eight sets of 20-second high-effort exercises with 30-second rest intervals, totaling 370 seconds of activity. The primary metrics evaluated were blood lactate levels, heart rate (HR), rating of perceived exertion (RPE), and training impulse (TRIMP). Participants in the enzyme group received a fruit and vegetable enzyme supplement in a 30 c.c. dose twice daily for 14 days. The study aimed to determine if enzyme supplementation could effectively mitigate the physiological stress of HIIE and improve exercise outcomes in the elderly.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 65 and above
2. healthy elderly participants
3. regular exercise habit (3 times per week within the past year)
4. Those who can move their upper and lower limbs normally

Exclusion Criteria:

1. no history of upper limb skeletal muscle injury or major injury
2. No heart-related diseases such as high blood pressure
3. No related chronic diseases, such as diabetes

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-25 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Lactate | pre and after-intervention: measurements taken before the test, during the 2 and 4 minute of the test, and 5 and 10 minutes after the test.
  Measure lactate level with fingertip blood test in Exergaming HIIE
Heart rate (bpm) | Collect the heart rate at 20, 50, 80, 110, 140, 170, 200 and 220 seconds in the HIIE test
  Use a heart rate monitor to record heart rate in Exergaming HIIE
Borg 0-10 score rating of perceived exertion (RPE) | Collect the RPE at 20, 50, 80, 110, 140, 170, 200 and 220 seconds in the HIIE test
  Use Borg 0-10 score RPE to record RPE in Exergaming HIIE

SECONDARY OUTCOMES:
Training Impulse | During Exergaming HIIE
  Calculate the subjective and objective training Impulse (arbitrary unit, AU) based on the heart rate and RPE.

CONTACTS AND LOCATIONS:
Locations (1):
- Tainan University of Technology, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-15): https://cdn.clinicaltrials.gov/large-docs/08/NCT06466408/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-15): https://cdn.clinicaltrials.gov/large-docs/08/NCT06466408/ICF_001.pdf